CLINICAL TRIAL: NCT05600803
Title: Efficacy of Single-operator Cholangioscopy to Screen for Neoplastic Bile Duct Lesions in Patients With Bile Duct Stones
Brief Title: Screening Single-operator Cholangioscopy for Neoplastic Bile Duct Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong Ho Moon, MD, PhD, FASGE, FJGES, Soonchunhyang University Hospital
Other Study IDs: screeningsoc
Record Dates: First submitted 2022-10-26; First posted 2022-11-01 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Cholangiocarcinoma; Bile Duct Neoplasms
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DSOC group: Study subjects are patients who satisfied the inclusion/exclusion criteria and underwent single-operator cholangioscopy.
  Interventions: Procedure: Single-operator cholangioscopy

INTERVENTIONS:
Procedure: Single-operator cholangioscopy — SpyGlass (Boston Scientific Co, Marlborough, USA) which enabled the direct visualization of the pancreaticobiliary system for the evaluation of intraductal lesions

SUMMARY:
This is the prospective observational study to explore whether the SpyGlass DS II system could be used to screen early-stage neoplastic bile duct lesions in selected patients.

DETAILED DESCRIPTION:
It is difficult to diagnose neoplastic bile duct lesions (including cholangiocarcinomas) via direct endoscopic evaluation of the bile duct. Most evaluations of biliary lesions have used indirect imaging modalities such as CT, MRI, or ERCP. However, CT and MRI do not yield tissue diagnoses, unlike ERCP, although the diagnostic accuracy for the latter remains unsatisfactory. Recently, remarkable advances in cholangioscopic systems have been made. Of the currently available cholangioscopic systems, the SpyGlass (Boston Scientific Co, Natick, Mass, USA) is a disposable cholangioscope permitting 4-way deflected steering by a single operator. We aimed to evaluate the efficacy of single-operator cholangioscopy (SpyGlass DS II system) to screen for neoplastic bile duct lesions in patients with bile duct stones, which is one of the risk factor of cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 18 years
2. Patients with risk factors for CCA (viral hepatitis, parasitic infection, choledochal cyst, primary sclerosing cholangitis, biliary stones, and toxins)
3. Patients who undergo ERCP for confirmation of CBD clearance
4. Dilated common bile duct (> 10 mm)
5. Previous sphincteroplasty, such as major endoscopic sphincterotomy and/or endoscopic papillary balloon dilatation

Exclusion Criteria:

1. Presence of biliary tract cancer
2. Presence of distal CBD stricture
3. Bleeding tendency (INR>1.5 or platelets <50000 mm3)
4. Contraindications of ERCP

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to recruit a total of 239 patients, assuming that the detection rate of neoplastic bile duct is about 3.5% by referring to the preceding literature. (one-sample inference for binomial proportions, one-sided test, significance 5%, power 80%)
Sampling Method: Non-Probability Sample
Enrollment: 236 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
detection rate | Until the end of the single-operator cholangioscopy session (up to 20 minutes)
  detection rate of intraductal neoplastic lesions in patients with bile duct stones who underwent single-operator cholangioscopy

SECONDARY OUTCOMES:
Technical success of cholangioscopy | Up to 15 minutes from the time the endoscope passes through the oral cavity
  successful insertion of the cholangioscope through the ampulla of Vater and advancement up to the bifurcation of the biliary tree
Technical success of cholangioscopy-guided biopsy | Until the end of the single-operator cholangioscopy session (up to 20 minutes)
  successful tissue sampling of intraductal superficial lesions under direct visualization
Adverse events | From the start of endoscopy to the end of the study observation period (at least 12 months)
  all adverse events including cholangitis, pancreatitis, perforation, bleeding, and air embolism based on ASGE criteria
Number needed to screen | From the start of endoscopy to the end of the study observation period (at least 12 months)
  the number of persons who would need to be screened to diagnose one neoplastic bile duct lesion in selected patients

CONTACTS AND LOCATIONS:
Locations (1):
- Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
By sharing and conducting research, we try to share pain and optimize performance through cooperation. Details have not been decided yet.

REFERENCES:
- [Background] Moon JH, Terheggen G, Choi HJ, Neuhaus H. Peroral cholangioscopy: diagnostic and therapeutic applications. Gastroenterology. 2013 Feb;144(2):276-282. doi: 10.1053/j.gastro.2012.10.045. Epub 2012 Nov 2. No abstract available. PMID 23127575
- [Background] Siddiqui AA, Mehendiratta V, Jackson W, Loren DE, Kowalski TE, Eloubeidi MA. Identification of cholangiocarcinoma by using the Spyglass Spyscope system for peroral cholangioscopy and biopsy collection. Clin Gastroenterol Hepatol. 2012 May;10(5):466-71; quiz e48. doi: 10.1016/j.cgh.2011.12.021. Epub 2011 Dec 16. PMID 22178463
- [Background] Chen YK, Parsi MA, Binmoeller KF, Hawes RH, Pleskow DK, Slivka A, Haluszka O, Petersen BT, Sherman S, Deviere J, Meisner S, Stevens PD, Costamagna G, Ponchon T, Peetermans JA, Neuhaus H. Single-operator cholangioscopy in patients requiring evaluation of bile duct disease or therapy of biliary stones (with videos). Gastrointest Endosc. 2011 Oct;74(4):805-14. doi: 10.1016/j.gie.2011.04.016. Epub 2011 Jul 18. PMID 21762903
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Imperiale TF, Wagner DR, Lin CY, Larkin GN, Rogge JD, Ransohoff DF. Results of screening colonoscopy among persons 40 to 49 years of age. N Engl J Med. 2002 Jun 6;346(23):1781-5. doi: 10.1056/NEJM200206063462304. PMID 12050337
- [Background] Saraiva MM, Ribeiro T, Ferreira JPS, Boas FV, Afonso J, Santos AL, Parente MPL, Jorge RN, Pereira P, Macedo G. Artificial intelligence for automatic diagnosis of biliary stricture malignancy status in single-operator cholangioscopy: a pilot study. Gastrointest Endosc. 2022 Feb;95(2):339-348. doi: 10.1016/j.gie.2021.08.027. Epub 2021 Sep 8. PMID 34508767
- [Result] Shin IS, Moon JH, Lee YN, Kim HK, Lee TH, Yang JK, Cha SW, Cho YD, Park SH. Use of peroral cholangioscopy to screen for neoplastic bile duct lesions in patients with bile duct stones (with videos). Gastrointest Endosc. 2021 Oct;94(4):776-785. doi: 10.1016/j.gie.2021.03.997. Epub 2021 Apr 15. PMID 33865838